CLINICAL TRIAL: NCT04812327
Title: Capturing Infectious COVID-19 Asymptomatic Cases in Singapore
Status: Withdrawn | Type: Observational
Why Stopped: Study was cancelled prior enrollment due to business decision.
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: SGP-21AsymVer-01
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Covid19; SARS CoV-2
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Observational Diagnostic Evaluation: Potential participants will be recruited at study sites where they are admitted/held for COVID-19 isolation. On the first day of isolation (ideally on the day they first test positive for SARS-CoV-2), potential participants will be asked to participate in the study. After consent (Study Day 0), two nasopharyngeal swabs (NP swabs) and one nasal swab will be collected. One NP swab will be tested via viral culture and the other nasal swab will be tested by RT-PCR for SARS-CoV-2. The nasal swab will be tested on the BD Veritor System. Specimen collection and testing will be repeated every 2 days for 6 days (Study Day 2, Day 4, and Day 6) or until the RT-PCR Ct value is >30, whichever comes first. Participants will be monitored for symptoms of COVID-19 throughout the study.
  Interventions: Diagnostic Test: BD Veritor Plus System for Rapid Detection of SARS CoV-2; Diagnostic Test: rt-PCR; Diagnostic Test: viral culture

INTERVENTIONS:
Diagnostic Test: BD Veritor Plus System for Rapid Detection of SARS CoV-2 — Nasal Sawb for the conduct of the Veritor Antigen Test
Diagnostic Test: rt-PCR — Nasopharyngeal Swab for the conduct of a rt-PCR
Diagnostic Test: viral culture — Nasopharyngeal Swab for the conduct of viral culture

SUMMARY:
This study is being conducted to assess the performance of the BD Veritor™ Plus System for Rapid Detection of SARS-CoV-2, used in serial testing, in identification of infectious, asymptomatic individuals. This information may be used to inform development of an effective testing strategy by policy makers.

DETAILED DESCRIPTION:
This multi-center, prospective, observational, diagnostic evaluation study is designed to assess the performance of the BD Veritor System in the detection of SARS-CoV-2 in asymptomatic individuals compared to viral culture and a commercially available RT-PCR assay over multiple testing time points. The study will enroll a minimum of 150 asymptomatic, adult participants who test positive for SARS-CoV-2 during community/traveler screening procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥21 years of age at the time of informed consent
2. Has a positive screening test for SARS-CoV-2 by RT-PCR
3. Is asymptomatic for COVID-19 on the day of their positive screening test (may have symptoms on the actual day of study enrollment)
4. Is expected to remain at the study site for the full 6-day study period
5. Willing and able to complete all study required procedures
6. Provision of signed and dated informed consent form

Exclusion Criteria:

1. History of frequent or difficult to control nosebleeds within the 14 days prior to study participation
2. If, at the discretion of the Investigator, involvement in the study is likely to jeopardize the subject's health or their current or future medical treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at study sites from individuals admitted for SARS-CoV-2 isolation. Once enrolled, participants may be transferred to a different care unit, or units, throughout their time in the study depending on their medical needs.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Assess the performance of the BD Veritor System for Rapid Detection of SARS-CoV-2 compared viral culture, over multiple collection time points | 6 days
  * Assay results: Positive percent agreement (PPA)
  * Assay results: Negative percent agreement (NPA)

SECONDARY OUTCOMES:
Assess the performance of the BD Veritor System for Rapid Detection of SARS-CoV-2 compared to a commercially available RT-PCR asay, over multiple collection time points | 6 days
  * Assay results: Positive percent agreement (PPA)
  * Assay results: Negative percent agreement (NPA)
Assess the performance a commercially available RT-PCR assay compared to viral culture, over multiple test time points | 6 days
  * Assay results: Positive percent agreement (PPA)
  * Assay results: Negative percent agreement (NPA)

CONTACTS AND LOCATIONS:
Overall Officials: Yen Seow Tan, MD, Principal Investigator — Hospital Employee
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No